CLINICAL TRIAL: NCT05343468
Title: Independence, Quality of Life, and Adaptive Behavioral Skills Improved in Children With Down Syndrome After Using Assistive Technology
Brief Title: Life Skills Improved in Children With Down Syndrome After Using Assistive Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MapHabit, Inc. (Industry)
Collaborators: LuMind IDSC Foundation (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Stuart Zola, Chief Scientific Officer, MapHabit, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LuMind Study; 5R43AG065081-02 (NIH)
Record Dates: First submitted 2022-04-05; First posted 2022-04-25 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Down Syndrome; Adaptive Behavior; Quality of Life
Keywords: Down syndrome; Assistive technology; Adaptive behavioral skills
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Intervention Model Description: This single-arm repeated measures design examined the effects of a software device as an intervention, permitting the participants to serve as their own controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): Singe-arm: the assistive digital software was implemented as an intervention to all participants.
  Interventions: Device: The MapHabit System

INTERVENTIONS:
Device: The MapHabit System — The MapHabit System (MHS) is a commercially available visual mapping software application that utilize visual, audio, and text media to create step-by-step visual guides to assist individuals and their caregivers in structuring and accomplishing activities of daily living (ADLs). The goal of the application is to develop and facilitate habits and routines using structured visual and auditory stimuli that can be customized by the user and can include educational and lesson-based material in addition to ADLs. The application was made available to families through compatible smartphones and tablets.
  The MHS is a general wellness product and there is no regulatory oversight of the MapHabit System mapping functionality. This functionality is not a regulated medical device.

SUMMARY:
Enhancing independence and quality of life are key modifiable outcomes that are short- and long-term goals for children with Down syndrome (DS) and for their parents. The study investigated the efficacy of assistive technology in improving children with Down Syndrome's independence and quality of life. Using a commercially available assistive technology, the MapHabit system, the investigators implemented the software with participants' families for 4 weeks. The investigators hypothesized that the assistive technology will improve adaptive behavioral skills and overall quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Down syndrome diagnosis
* Age between 7-17
* Internet access
* Proficiency in English

Exclusion Criteria:

* Ages outside of 7-17
* Located outside of the United States of America
* No internet access
* No proficiency in English

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2020-09-20 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-08-05 (Actual)

PRIMARY OUTCOMES:
Change in Adaptive Behavior Assessment System Third Edition (ABAS-3) from Baseline at 4 Weeks | Pre-Post: The assessment was administered at the beginning and end of the study's duration (4-week study).
  Assessment is used commonly for children with Down syndrome that evaluates conceptual, social, and practical behavioral skills that are significant for day-to-day functioning. The assessment is scored with the General Adaptive Composite (GAC), which summarizes performance across all adaptive skill areas. GAC score ranges from 0-130, with a higher score indicating better outcome.
Quality of Life - 18 (QoL-18) | The instrument was administered to the participants after the completion of the study duration (4-week study).
  18-item quality-of-life questionnaire (QoL-18) evaluated a range of participants' behaviors, including mood, engagement, and memory at the end of the study compared to before the use of the MHS. The instrument is scored on a Likert Scale, ranging from 1-5. A higher number indicates better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Zola, PhD, Principal Investigator — MapHabit, Inc.
Locations (1):
- MapHabit, Inc., Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal. Proposals should be directed to szola@maphabit.com. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Boatman F, Golden M, Jin J, Kim Y, Law S, Lu A, Merriam N, Zola S. Assistive technology: Visual mapping combined with mobile software can enhance quality of life and ability to carry out activities of daily living in individuals with impaired memory. Technol Health Care. 2020;28(2):121-128. doi: 10.3233/THC-191980. PMID 31796718
- [Background] Kelleher J, Zola S, Cui X, Chen S, Gerber C, Parker MW, Davis C, Law S, Golden M, Vaughan CP. Personalized Visual Mapping Assistive Technology to Improve Functional Ability in Persons With Dementia: Feasibility Cohort Study. JMIR Aging. 2021 Oct 19;4(4):e28165. doi: 10.2196/28165. PMID 34269690
- [Background] Parker MW, Davis C, White K, Johnson D, Golden M, Zola S. Reduced care burden and improved quality of life in African American family caregivers: Positive impact of personalized assistive technology. Technol Health Care. 2022;30(2):379-387. doi: 10.3233/THC-213049. PMID 34334439
- [Derived] White K, Han SS, Britton A, Hendrix J. A feasibility study demonstrating that independence, quality of life, and adaptive behavioral skills can improve in children with Down syndrome after using assistive technology. PLoS One. 2023 May 24;18(5):e0284738. doi: 10.1371/journal.pone.0284738. eCollection 2023. PMID 37224142